CLINICAL TRIAL: NCT04434170
Title: Valutazione Della capacità d'Esercizio, Della funzionalità Respiratoria e Del Rimodellamento Ventricolare Sinistro in Pazienti Affetti da Scompenso Cardiaco a Frazione d'Eiezione Ridotta Trattati Con Sacubitril/Valsartan
Brief Title: Effects of Sacubitril/Valsartan on Exercise Capacity, Natriuretic Peptides and Ventricular Remodeling in Heart Failure
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, Prof, Centro Cardiologico Monzino
Other Study IDs: Entresto CPET
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: sacubitril/valsartan; exercise; cardiopulmonary exercise test; left ventricular remodeling
MeSH Terms: conditions — Heart Failure; Motor Activity; Ventricular Remodeling | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart failure: outpatients with heart failure with reduced ejection fraction in treatment with sacubitril/valsartan according to guidelines
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — outpatients who start treatment with sacubitril/valsartan according to guidelines will andergo cardiopulmonary exercise testing evaluation

SUMMARY:
Background: Sacubitril/valsartan, a novel therapy in the treatment of heart failure with reduced ejection fraction (HFrEF), has recently proved efficacy in improving exercise tolerance and cardiac performance. Cardiopulmonary exercise test (CPET) provides functional prognostic parameters for patient with HFrEF (i.e. peakVO2 and ventilation/CO2 production [VE/VCO2] slope) and it is a well-recognized, valuable, accurate tool for risk stratification.

Aim of the study and methods: The aim of the study is to prospectively enroll a cohort of 100 HFrEF outpatients eligible for sacubitril/valsartan and perform serial CPET, laboratory and echocardiographic assessments before and during the gradual titration of the treatment, in order to evaluate its effects on cardiopulmonary function and left ventricular remodeling. The procedures will be repeated along the follow-up at 1, 2 and 3 months after the enrollment (titration period) and at 6 months after the reach of the maximum tolerated dose.

DETAILED DESCRIPTION:
Given the recent introduction of the drug into the clinical routine, the evaluation of the experience "on the field" is important to refine the clinical management of patients treated with sacubitril / valsartan. Furthermore, at the moment sacubitril / valsartan has proven effective in some small preliminary studies in improving the ejection fraction and some echocardiographic parameters of ventricular remodeling on top of the concomitant optimal medical therapy, although further data are needed in this regard.

In particular, the potential benefits on exercise capacity, respiratory function parameters and left ventricular remodeling in heart failure patients treated with sacubitril / valsartan has not been studied extensively at the moment. In this regard, the cardiopulmonary exercise test (CPET) allows to obtain prognostic functional parameters in patients with chronic heart failure such as peak V02 (peak V02) and the ventilation / production of C02 slope (VE / VC02 slope). CPET is a valid, recognized and accurate tool for risk stratification in heart failure patients.

Furthermore, few data are available on lung diffusion (DLCO) and on specific markers of the alveolar-capillary membrane, such as type B surfactant proteins (SPB) in patients treated with sacubtril / valsartan. Our team has already shown how these biomarkers and DLCO are influenced by drug treatments such as Levosimendan and Ace inhibitors.

The aim of the study is to evaluate the exercise capacity, spirometry, echocardiographic parameters of left ventricular sistolic and diastolic function, Nt-proBNP dosage and quality of life and the related dose-effect correlation in a multicenter cohort of 100 patients with stable heart failure (class functional NYHA II e lII) and reduced left ventricular ejection fraction in patients eligible for sacubitril / valsartan treatment.

A subgroup of patients will be also analyzed for data relating to the effect of sacubitril / valsartan on DLCO and blood levels of Surfactant Bindig protein (SPB).

Sacubitril / Valsartan will be prescribed according to guidelines, initially at the lowest dosage of 24/26 mg b.i.d. to verify its tolerability with the prospect of gradually increasing the dosage during subsequent follow-up visits. The re-evaluation of the treatment and the titration of the sacubitril / valsartan dose will take place every 4 weeks until the maximum tolerated dose is reached. The dose under study will be the maximum tolerated by the patient (however not higher than 97 mg / 103mg bd).

Cardiological examination with ECG, spirometry, CPET, the Kansas City Cardiomyopathy Questionnaire, blood count, creatinine, nitrogen, sodium, potassium, chlorine and NTproBNP will be performed at each visit (from Baseline to 6 months). The colordoppler echocardiogram will instead be performed only at the baseline and after 6 months.

A subset of patients will also be subjected to analysis of the blood levels of SPB and DLCO at baseline and 6 months after reaching the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class (NYHA) II-III
* stable clinical conditions
* reduced ejection fraction (< 35%)
* capability to perform a cardiopulmonary exercise test (CPET)

Exclusion Criteria:

* moderate-severe chronic obstructive pulmonary disease
* chronic oxygen therapy
* contraindication to CPET
* planned procedures (i.e. cardiac surgery, revascularization procedures, CRT implantation) that could per se impact on CPET, echocardiography and laboratory values

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HFrEF outpatients eligible for sacubitril/valsartan according to guidelines and perform serial CPET, laboratory and echocardiographic assessments before and during the gradual titration of the treatment
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
VO2 evaluation after treatment | 1 month after start of treatment with sacubitril/valsartan
  changes in peak VO2 at cardiopulmonary exercise test
VO2 evaluation after treatment | 2 months after start of treatment with sacubitril/valsartan
  changes in peak VO2 at cardiopulmonary exercise test
VO2 evaluation after treatment | 3 months after start of treatment with sacubitril/valsartan
  changes in peak VO2 at cardiopulmonary exercise test
VO2 evaluation after treatment | 9 months after start of treatment with sacubitril/valsartan
  changes in peak VO2 at cardiopulmonary exercise test

SECONDARY OUTCOMES:
lung function evaluation after treatment | 1 month after start of treatment with sacubitril/valsartan
  changes in FVC, FEV1, PEF and FEV1%, by spirometry
lung function evaluation after treatment | 2 months after start of treatment with sacubitril/valsartan
  changes in FVC, FEV1, PEF and FEV1%, by spirometry
lung function evaluation after treatment | 3 months after start of treatment with sacubitril/valsartan
  changes in FVC, FEV1, PEF and FEV1%, by spirometry
lung function evaluation after treatment | 9 months after start of treatment with sacubitril/valsartan
  changes in FVC, FEV1, PEF and FEV1%, by spirometry
DLCO | 1 month after start of treatment with sacubitril/valsartan
  DLCO evaluation
DLCO | 9 months after start of treatment with sacubitril/valsartan
  DLCO evaluation
Surfactant B-type protein after treatment | 1 month after start of treatment with sacubitril/valsartan
  SPB quantification
Surfactant B-type protein after treatment | 9 months after start of treatment with sacubitril/valsartan
  SPB quantification
left ventricular remodeling | 1 month after start of treatment with sacubitril/valsartan
  ejection fraction
left ventricular remodeling | 2 months after start of treatment with sacubitril/valsartan
  ejection fraction
left ventricular remodeling | 9 months after start of treatment with sacubitril/valsartan
  ejection fraction
left ventricular remodeling | 1 month after start of treatment with sacubitril/valsartan
  End-diastolic and end-systolic left ventricular volumes
left ventricular remodeling | 2 months after start of treatment with sacubitril/valsartan
  End-diastolic and end-systolic left ventricular volumes
left ventricular remodeling | 9 months after start of treatment with sacubitril/valsartan
  End-diastolic and end-systolic left ventricular volumes

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided